CLINICAL TRIAL: NCT00027937
Title: A Phase II Study Of Mobilization Chemotherapy With GMCSF And GCSF Followed By High Dose Therapy Combined With IL2 Activated Autologous Peripheral Blood Stem Cells Followed By Sequential IL2 Therapy As Treatment For Solid Tumors And Lymphoma
Brief Title: Combination Chemotherapy, Peripheral Stem Cell Transplantation, and Biological Therapy in Treating Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1595.00; FHCRC-1595.00; IMMUNEX-FHCRC-1595.00; NCI-G01-2037; CDR0000069095 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aldesleukin; Filgrastim; sargramostim; Busulfan; Cyclophosphamide; Melphalan; Paclitaxel; Thiotepa

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: sargramostim
Drug: busulfan
Drug: cyclophosphamide
Drug: melphalan
Drug: paclitaxel
Drug: thiotepa
Procedure: bone marrow ablation with stem cell support
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Biological therapies such as interleukin-2 use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, peripheral stem cell transplantation, and interleukin-2 in treating patients who have solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of sargramostim (GM-CSF) and filgrastim (G-CSF)-mobilized interleukin-2(IL-2)-incubated autologous peripheral blood stem cells and sequential IL-2 in patients with solid tumors or lymphoma.
* Determine the ability of cyclophosphamide and paclitaxel followed by GM-CSF and G-CSF to mobilize adequate numbers of CD34+ cells and immune cells in these patients.
* Determine the time to neutrophil and platelet engraftment in patients treated with this regimen.
* Determine the overall and disease-free survival of patients treated with this regimen.

OUTLINE: Patients receive cyclophosphamide IV over 1-2 hours on day 1 and paclitaxel IV over 4 hours on day 2. Patients also receive sargramostim (GM-CSF) subcutaneously (SC) alone on days 3-9 and GM-CSF and filgrastim (G-CSF) SC beginning on day 10 and continuing until leukapheresis is completed.

Patients receive high-dose chemotherapy comprising oral busulfan every 6 hours on days -8 to -6, melphalan IV on days -5 and -4, and thiotepa IV on days -3 and -2. Autologous peripheral blood stem cells (PBSC) are treated ex vivo with interleukin-2 (IL-2) on day -1. Patients undergo IL-2-treated autologous PBSC transplantation on day 0.

Beginning 4 hours after PBSC transplantation, patients receive IL-2 IV continuously for 5 days. IL-2 therapy repeats every 7 days for 4 courses.

Patients are followed on days 60-80, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor, Hodgkin's lymphoma, or B-cell non-Hodgkin's lymphoma
* Eligible for autologous stem cell transplantation
* No pleural effusion, pericardial effusion, or ascites
* No T-cell lymphoma

PATIENT CHARACTERISTICS:

Age:

* Under 57

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 mg/dL (unless due to Gilbert's disease)
* SGOT or SGPT no greater than 2 times upper limit of normal
* Hepatitis B and C negative

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* LVEF at least 50%
* No congestive heart disease
* No history of myocardial infarction within the past year
* No coronary artery disease
* No history of arrhythmia

Pulmonary:

* Diffusion capacity (corrected) at least 60%
* FEV_1 at least 65% of predicted

Other:

* HIV negative
* No history of seizures
* No mental disorders requiring medication (e.g., haloperidol)
* No active connective tissue disease
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or any carcinoma in situ
* No allergy to gentamicin
* No hypersensitivity to E. coli-derived preparations
* No history of severe allergy to sargramostim (GM-CSF) or filgrastim (G-CSF)
* No systemic infection
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent corticosteroid therapy

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No contrast dye for 3 weeks after completion of interleukin-2 therapy

Max Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2001-08; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States